CLINICAL TRIAL: NCT01486862
Title: NovoMix® 30 (Biphasic Insulin Aspart 70/30) Titrate-to-target: An Observational Study of the Efficacy of NovoMix® 30 in Subjects With Type 2 Diabetes Mellitus Not Achieving Glycaemic Targets on OADs
Brief Title: Efficacy of Biphasic Insulin Aspart 30 in Subjects With Type 2 Diabetes Failing on OADs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1673
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIAsp 30 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Dose individually adjusted. Administered once daily for 16 weeks. If HbA1c after 16 weeks of treatment is above 7.0%, insulin is administered twice daily for additional 16 weeks.

SUMMARY:
This trial is conducted in North America. The aim of this trial is to investigate the efficacy of biphasic insulin aspart 30 in subjects with type 2 diabetes not achieving glycaemic targets on OADs (oral anti-diabetic drugs).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus for at least 12 months
* HbA1c between 7.5-14.5% (inclusive) at screening
* Insulin naïve
* An antidiabetic regimen that has been stable for at least 3 months prior to screening
* An antidiabetic regimen that includes a minimum of 2 OADs

Exclusion Criteria:

* Use of any insulin preparations within the past 6 months
* Active proliferative retinopathy or maculopathy requiring treatment within 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving HbA1c (glycosylated haemoglobin A1c) below 7.0%

SECONDARY OUTCOMES:
Change in HbA1c
Total number of hypoglycemic events
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Pachuca, Mexico

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com